CLINICAL TRIAL: NCT05273047
Title: Assessment and Follow-up of Patients With KRAS G12C-mutated Metastatic Non-Small Cell Lung Cancer Who Received Sotorasib as Part of the French Early Access Program (ATU)
Brief Title: RW Efficacy of Sotorasib in KRAS G12C-mutated Metastatic NSCLC
Acronym: LungKG12Ci
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: IFCT-2102
Record Dates: First submitted 2022-02-24; First posted 2022-03-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Nsclc; KRAS P.G12C
Keywords: sotorasib; real-world study; KRAS P.G12C; NSCLC; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the IFCT2102 Lung KG12Ci study is to closely monitor cohort ATU applications in order to collect retrospectively, as soon as possible after inclusion and under real-life conditions, the efficacy data on sotorasib (AMG 510) as well as the demographic and molecular characteristics of patients.

DETAILED DESCRIPTION:
The purpose of the IFCT2102 Lung KG12Ci study is to closely monitor cohort ATU applications in order to collect retrospectively, as soon as possible after inclusion and under real-life conditions, the efficacy data on sotorasib (AMG 510) as well as the demographic and molecular characteristics of patients.

The objective of this retrospective observational, multicenter, cohort study is to describe, in real life, the characteristics and evolution of NSCLC patients with a KRAS G12C mutation, treated with sotorasib in the framework of the cohort ATU in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage IV NSCLC at time of initiation of treatment with sotorasib
* Presence of KRAS G12C mutation diagnosed on tumor sample and/or on liquid biopsy (co mutations allowed)
* Patients who received at least one dose of the treatment with sotorasib as part of the French Early Access Program (ATU program)
* Patients who were informed about the study and do not object for their data to be collected
* Age > 18 years

Exclusion Criteria:

* Patients enrolled in a sotorasib clinical trial
* Patients with a psychiatric history that hinders the comprehension of the information leaflet
* Patients under curatorship or guardianship
* Unable to obtain data collection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic Non-Small Cell Lung Cancer (NSCLC) harboring KRAS G12C mutation who received sotorasib as second line treatment or more as part of the French Early Access Program (ATU program).
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Real-world progression-free survival (rwPFS) | through study completion, an average of 1.5 year
  rwPFS will be defined as the time from the date of the first dose of treatment with sotorasib to the date of first occurrence of disease progression (defined by the treating physician) or death from any cause during the study
Patients' clinical and biological characteristics at NSCLC diagnosis and initiation of sotorasib | 6 months
  Stage cTNM, smoking habits, PS, presence of brain metastasis, gender, age, histological, KRAS and other biomarkers status
Overall survival (OS) | through study completion, an average of 1.5 year
  OS will be determined as the time from the date of first dose of treatment with sotorasib to the date of death due to any cause during the study
Duration of treatment with sotorasib | through study completion, an average of 1.5 year
  Duration of treatment is defined as the time from the date of first dose of treatment with sotorasib to the date of discontinuation of treatment with sotorasib or death from any cause during the study
Best response (complete response, partial response, stable disease, progression) | through study completion, an average of 1.5 year
  Best response will be defined as the best response recorded from the start of treatment with sotorasib until disease progression or start of further anti-cancer treatment
Duration of response | through study completion, an average of 1.5 year
  Duration of response will be defined as the time from the date of the first documented response (complete or partial) to the earliest date of disease progression
Duration of treatment with sotorasib beyond 1rst progression | through study completion, an average of 1.5 year
  Duration of treatment with sotorasib beyond progression will be defined as time between first occurrence of disease progression and treatment discontinuation
Description of treatments received before and after sotorasib treatment | through study completion, an average of 1.5 year
  Description of treatments received before and after sotorasib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Céline Mascaux, Study Chair — Strasbourg - CHU; Florian Guisier, Study Chair — Rouen - CHU
Locations (3):
- France (3):
  - Paris - Hôpital Cochin, Paris
  - Rouen - CHU, Rouen
  - Strasbourg - CHU, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/803-ifct-2102